CLINICAL TRIAL: NCT00932360
Title: Transcutaneous Electrical Nerve Stimulation (TENS) and Fibromyalgia (FM)
Acronym: TENS&FM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana Dailey (Other)
Collaborators: American Physical Therapy Association (Other)
Responsible Party: Sponsor-Investigator, Dana Dailey, Research Associate, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 200903744; NCT00750321 (obsolete NCT alias)
Record Dates: First submitted 2009-06-23; First posted 2009-07-03 (Estimated); Results first posted 2019-01-10 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Transcutaneous Electrical Nerve Stimulation (TENS)
MeSH Terms: conditions — Fibromyalgia | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (6):
- Active TENS Placebo TENS No TENS (Experimental): Active TENS: 100 Hz, 200 μs at maximal tolerable intensity Placebo TENS: 100 Hz, 200 μs on for 45 seconds and then ramped off No TENS: Participants wore a TENS unit that was turned off for blinding of the outcome assessor
  Interventions: Device: TENS
- Placebo TENS Active TENS No TENS (Experimental): Placebo TENS: 100 Hz, 200 μs on for 45 seconds and then ramped off Active TENS: 100 Hz, 200 μs at maximal tolerable intensity Participants wore a TENS unit that was turned off for blinding of the outcome assessor
  Interventions: Device: TENS
- No TENS Active TENS Placebo TENS (Experimental): No TENS: Participants wore a TENS unit that was turned off for blinding of the outcome assessor Active TENS: 100 Hz, 200 μs at maximal tolerable intensity Placebo TENS: 100 Hz, 200 μs on for 45 seconds and then ramped off
  Interventions: Device: TENS
- Active TENS No TENS Placebo TENS (Experimental): Active TENS: 100 Hz, 200 μs at maximal tolerable intensity No TENS: Participants wore a TENS unit that was turned off for blinding of the outcome assessor Placebo TENS: 100 Hz, 200 μs on for 45 seconds and then ramped off
  Interventions: Device: TENS
- Placebo TENS No TENS Active TENS (Experimental): Placebo TENS: 100 Hz, 200 μs on for 45 seconds and then ramped off Participants wore a TENS unit that was turned off for blinding of the outcome assessor Active TENS: 100 Hz, 200 μs at maximal tolerable intensity
  Interventions: Device: TENS
- No TENS Placebo TENS Active TENS (Experimental): No TENS: Participants wore a TENS unit that was turned off for blinding of the outcome assessor Placebo TENS: 100 Hz, 200 μs on for 45 seconds and then ramped off Active TENS: 100 Hz, 200 μs at maximal tolerable intensity
  Interventions: Device: TENS

INTERVENTIONS:
Device: TENS — Active TENS, Placebo TENS and No Treatment TENS
  Other Names: Rehabilicare Maxima

SUMMARY:
Fibromyalgia as a clinical syndrome is defined by chronic widespread muscular pain, fatigue and tenderness with hyperalgesia to pressure over tender points. Pain associated with fibromyalgia can interfere with daily function, work, and social activities. Thus, one of the main treatments for patients with fibromyalgia must focus on pain relief to allow the person to function more independently both at home and at work. Although the etiology of fibromyalgia is unknown, there is clearly enhanced sensitization in the central nervous system pain pathways as demonstrating by decreases in pressure pain thresholds, reduced central inhibition, and enhanced temporal summation. Reducing pain in people with fibromyalgia would help increase the patient's ability to return to work, perform activities of daily living and thus improve the quality of life for the patient. Transcutaneous electrical nerve stimulation (TENS) is a modality utilized in physical therapy that delivers electrical stimulation through the skin and is used for both acute and chronic pain. TENS works by reducing central excitability and increasing central inhibition. Thus, the investigators hypothesize that application of Transcutaneous Electrical Nerve Stimulation (TENS) to patients with Fibromyalgia (FM) will reduce pain, reduce central excitability by restoring diffuse noxious inhibitory controls (DNIC), and reduce temporal summation and that this decrease in pain and/or central excitability will improve function. The primary aim of the study is to test the effectiveness of TENS on pain and central excitability in a crossover design study for patients with Fibromyalgia with random assignment to three treatments: no treatment control, placebo TENS and active high frequency TENS. A secondary aim is to test the effect of decreased pain and central excitability on function in patients with Fibromyalgia.

DETAILED DESCRIPTION:
The study will be a simple crossover design with the following three treatments (1) active TENS, (2) placebo TENS or (3) no treatment control randomly assigned. Subjects will draw the order for treatments (A, B, and C) out of a bowl at the initial testing session. This will determine the order of the testing. Each subject will receive all 3 treatments in random order.

The following tools will be used to measure subject characteristics (Fibromyalgia Impact Questionnaire, Tampa Scale of Kinesiophobia), pain (McGill Pain Questionnaire and Visual Analogue Scale), central excitability (pressure pain thresholds, temporal summation and DNIC) and function (6 minute walk test, range of motion, sit to stand test).

ELIGIBILITY:
Inclusion Criteria:

* Fibromyalgia diagnosis by a physician
* History of cervical or lumbar pain

Exclusion Criteria:

* TENS use in the last 5 years
* Pacemaker
* No use of opioids

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2009-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dana L Dailey, PT,PhD, Principal Investigator — University of Iowa; Kathleen A Sluka, PhD, Study Chair — University of Iowa; Barbara Rakel, PhD, Study Chair — University of Iowa
Locations (1):
- University of Iowa - Physical Therapy and Rehabilitation Science, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No
See Publication listed for data

REFERENCES:
- [Result] Dailey DL, Rakel BA, Vance CGT, Liebano RE, Amrit AS, Bush HM, Lee KS, Lee JE, Sluka KA. Transcutaneous electrical nerve stimulation reduces pain, fatigue and hyperalgesia while restoring central inhibition in primary fibromyalgia. Pain. 2013 Nov;154(11):2554-2562. doi: 10.1016/j.pain.2013.07.043. Epub 2013 Jul 27. PMID 23900134
- See also: PubMed Link for full text article — https://www-ncbi-nlm-nih-gov.proxy.lib.uiowa.edu/pmc/articles/PMC3972497/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects (125) were screened for eligibility via telephone. 82 were excluded and 43 were consented and enrolled at the University of Iowa
Pre-assignment Details: 43 subjects were consented and enrolled to the cross over design study. Subjects were randomized to treatment group order after providing written consent. The three treatment groups for randomization order included: active TENS, placebo TENS and no treatment TENS.
Groups:
- Active TENS, Placebo TENS and No TENS; Active TENS No TENS Placebo TENS; Placebo TENS Active TENS No TENS; Placebo TENS No TENS Active TENS; No TENS Active TENS Placebo TENS; No TENS Placebo TENS Active TENS: Active TENS: 100 Hz, 200 μs at maximal tolerable intensity Placebo TENS:TENS at 100 Hz, 200 μs for 30 seconds and then the current ramped off over a 15 second time frame No TENS: Participants wore a TENS unit that was turned off for blinding of the outcome assessor
Period: 1: Visit 1/Week1
Arm/Group | Active TENS, Placebo TENS and No TENS | Active TENS No TENS Placebo TENS | Placebo TENS Active TENS No TENS | Placebo TENS No TENS Active TENS | No TENS Active TENS Placebo TENS | No TENS Placebo TENS Active TENS
Started | 10 | 6 | 3 | 13 | 4 | 7
Completed | 10 | 6 | 3 | 13 | 4 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout (One Week)
Arm/Group | Active TENS, Placebo TENS and No TENS | Active TENS No TENS Placebo TENS | Placebo TENS Active TENS No TENS | Placebo TENS No TENS Active TENS | No TENS Active TENS Placebo TENS | No TENS Placebo TENS Active TENS
Started | 10 | 6 | 3 | 13 | 4 | 7
Completed | 10 | 6 | 3 | 13 | 2 | 7
Not Completed | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 2 | 0
Period: Visit 2/Week 2
Arm/Group | Active TENS, Placebo TENS and No TENS | Active TENS No TENS Placebo TENS | Placebo TENS Active TENS No TENS | Placebo TENS No TENS Active TENS | No TENS Active TENS Placebo TENS | No TENS Placebo TENS Active TENS
Started | 10 | 6 | 3 | 13 | 2 | 7
Completed | 10 | 6 | 3 | 13 | 2 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout (One Week)
Arm/Group | Active TENS, Placebo TENS and No TENS | Active TENS No TENS Placebo TENS | Placebo TENS Active TENS No TENS | Placebo TENS No TENS Active TENS | No TENS Active TENS Placebo TENS | No TENS Placebo TENS Active TENS
Started | 10 | 6 | 3 | 13 | 2 | 7
Completed | 10 | 6 | 3 | 13 | 2 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Visit 3/Week 3
Arm/Group | Active TENS, Placebo TENS and No TENS | Active TENS No TENS Placebo TENS | Placebo TENS Active TENS No TENS | Placebo TENS No TENS Active TENS | No TENS Active TENS Placebo TENS | No TENS Placebo TENS Active TENS
Started | 10 | 6 | 3 | 13 | 2 | 7
Completed | 10 | 6 | 3 | 13 | 2 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: This is a crossover study with three groups. Subjects completed each arm of the study in random order.
Arm/Group | All Study Participants
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 42
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 42
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 2 subjects withdrew from the study after the first visit
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 43
    More than one race | 0
    Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants] — Population: 2 subjects withdrew after 1 visit
  participants
    United States | 43

OUTCOME MEASURES:

1. Primary Outcome: Pain at Rest Difference Score Pre-intervention and Post Intervention
Description: Visual Analog Scale 0-10 with 0 No Pain and 10 Worst Pain Imaginable Pain was measured at rest before and after intervention.
Time Frame: 3 weeks
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Active TENS; Placebo TENS; No TENS: Active and Placebo TENS with configured Rehabilicare Unit; No TENS with TENS worn and not turned on.
Arm/Group | Active TENS | Placebo TENS | No TENS
Number analyzed (Participants) | 43 | 43 | 41
units on a scale | 0.38 (0.26) | -0.74 (0.25) | -0.47 (0.26)

2. Primary Outcome: Pain With Movement Difference Score Pre-intervention and Post Intervention
Description: as for outcome 1
Time Frame: 3 weeks
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Active TENS to No Treatment to Placebo (ANP); Active TENS to Placebo to No Treatment (APN): Active and Placebo TENS with configured Rehabilicare Unit; No TENS with TENS worn and not turned on.
- No Treatment to Active TENS to Placebo TENS (NAP): Active and Placebo TENS with configured Rehabilicare Unit; No TENS with TENS worn and not turned on.r
Arm/Group | Active TENS to No Treatment to Placebo (ANP) | Active TENS to Placebo to No Treatment (APN) | No Treatment to Active TENS to Placebo TENS (NAP)
Number analyzed (Participants) | 43 | 43 | 41
score on a scale | 1.11 (0.26) | 0.23 (0.26) | 0.26 (0.25)

3. Secondary Outcome: Fatigue at Rest Difference Score Pre-intervention and Post Intervention
Description: Visual Analog Scale 0-10 with 0 No Fatigue and 10 Worst Fatigue Imaginable Pain was measured at rest before and after intervention.
Time Frame: 3 weeks
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Active TENS: 100 Hz, 200 μs at maximal tolerable intensity
- Placebo TENS: TENS at 100 Hz, 200 μs for 30 seconds and then the current ramped off over a 15 second time frame
- No TENS: Participants wore a TENS unit that was turned off for blinding of the outcome assessor
Arm/Group | Active TENS | Placebo TENS | No TENS
Number analyzed (Participants) | 43 | 43 | 41
units on a scale | -0.09 (0.21) | -0.14 (0.21) | 0.12 (0.22)

4. Secondary Outcome: Fatigue With Movement Difference Score Pre-intervention and Post Intervention
Description: as for outcome 3
Time Frame: 3 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Active TENS | Placebo TENS | No TENS
Number analyzed (Participants) | 43 | 43 | 41
units on a scale | 0.94 (0.23) | 0.39 (0.24) | 0.04 (0.23)

5. Secondary Outcome: PPT Cervical Region
Description: Pressure pain threshold cervical region (kPa)
Time Frame: 3 weeks
Measure: Mean (Standard Error); unit: pressure score (kPa)
Arm/Group | Active TENS | Placebo TENS | No TENS
Number analyzed (Participants) | 43 | 43 | 41
pressure score (kPa) | 53.15 (10.09) | 26.42 (10.02) | 19.39 (10.06)

6. Secondary Outcome: PPT Lumbar Region
Description: Pressure pain threshold in lumbar region (kPa)
Time Frame: 3 weeks
Measure: Mean (Standard Error); unit: pressure score (kPa)
Arm/Group | Active TENS | Placebo TENS | No TENS
Number analyzed (Participants) | 43 | 43 | 41
pressure score (kPa) | 86.97 (15.97) | 34.89 (15.91) | 33.23 (15.95)

7. Secondary Outcome: PPT for Anterior Tibialis
Description: Pressure pain threshold in leg (kPa)
Time Frame: 3 weeks
Measure: Mean (Standard Error); unit: pressure score (kPa)
Arm/Group | Active TENS | Placebo TENS | No TENS
Number analyzed (Participants) | 43 | 43 | 41
pressure score (kPa) | 62.86 (18.34) | 38.98 (21.85) | 4.4 (15.47)

8. Secondary Outcome: 6 Minute Walk Test Average Change (Feet)
Description: 6 minute walk test average change (feet) before and after intervention
Time Frame: 3 weeks
Measure: Mean (Standard Error); unit: feet
Arm/Group | Active TENS | Placebo TENS | No TENS
Number analyzed (Participants) | 43 | 43 | 41
feet | 41.85 (36.7) | -40.48 (36.31) | -0.97 (36.01)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Active TENS | Placebo TENS | No TENS
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/43 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/43 | 0/43
Other Adverse Events (participants affected / at risk) | 0/43 | 0/43 | 0/43

LIMITATIONS AND CAVEATS:
43 subjects were enrolled to the study and completed a treatment (Active TENS, Placebo TENS or No TENS) in a randomized order with a one week washout period between treatments. Results were analyzed by comparing the groups for outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes